CLINICAL TRIAL: NCT03568851
Title: Reproductive Health Outcomes by Method of Breast Milk Feeding
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Other Study IDs: 1198922
Record Dates: First submitted 2018-05-31; First posted 2018-06-26 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: Breast Feeding; Milk Expression, Breast; Amenorrhea, Postpartum
MeSH Terms: conditions — Breast Feeding; Breast Milk Expression; Amenorrhea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this research is to determine whether there are differences in ovarian suppression between women who are feeding at the breast compared with women who are pumping.

* In the main study, the aim is to compare reproductive health outcomes, including amenorrhea rates, duration of lactation, and resumption of sexual activity, between mothers who are exclusively breastfeeding (i.e. feeding at the breast) and those who are pumping after a term or preterm delivery.
* In the sub-study, the aim is to determine the feasibility and acceptability of using urinary luteinizing hormone (LH) detection kits at home to detect ovulation in exclusively breastmilk feeding women.

DETAILED DESCRIPTION:
Women will be recruited for this study during routine prenatal care. Interested and eligible participants will undergo an informed consent process. After, participants will answer questions regarding demographic information, medical history, obstetric and reproductive history, previous lactation history, and the Infant Feeding Intentions questionnaire.

Participants who are eligible after the second eligibility verification at the time of delivery hospitalization will be enrolled in the study. Enrolled participants will be given breastmilk and infant feeding logs to complete. Study staff will contact participants at 1, 2, 3, 4, 5, and 6 months after delivery to ask about breastmilk feeding practices in the last 24 hours, infant feeding, vaginal bleeding, sexual activity, use of contraceptive methods, and repeat pregnancies. In between the monthly phone calls, study staff will ask participants about the occurrence of vaginal bleeding.

For the sub-study, participants are recruited from the main study. Those who are eligible and interested will undergo an informed consent process. Participants will be given urinary LH detection kits and instructions for use at time of enrollment. Daily urine LH testing will start after 8 weeks postpartum. Participants will also receive monthly diaries to complete in addition to the breastmilk and infant feeding logs in the main study. Study staff will contact participants at 2, 3, 4, 5, and 6 months to review the diary information. If the urine LH test is positive, the participant will undergo a blood draw for serum progesterone levels to confirm ovulation.

The planned enrollment is 394 participants for the main study and 40 participants in the sub-study.

ELIGIBILITY:
MAIN STUDY

Inclusion Criteria:

* 15 through 45 years old
* planning to feeding her infant exclusively the mother's own milk for at least 6 months after delivery
* receiving prenatal care, plan to deliver, and plan to return to UC Davis for the postpartum visit
* 32 weeks gestation or greater at screening

Exclusion Criteria:

* have a multiple gestation pregnancy
* planning to initiate a hormonal contraceptive method at the postpartum visit

At time of delivery hospitalization, a second eligibility verification will occur and women will be excluded if they:

* initiated a hormonal contraceptive method (specifically intrauterine device, implant, depo provera injections) during the delivery hospitalization
* had a hysterectomy
* did not deliver at UC Davis
* are no longer interested in study participation

SUB-STUDY

Inclusion Criteria:

* enrolled in the main study
* within 8 weeks postpartum after delivering a singleton
* currently amenorrheic
* planning to continue breastmilk feeding for up to 6 months after delivery
* planning to avoid pregnancy in the first 6 months after delivery

Exclusion Criteria:

* less than 18 years old
* have a previous history of irregular or anovulatory cycles
* are using a hormonal method of contraception
* are unwilling to comply with study procedures

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Describes self as female
Study Population: Women who are planning on breastmilk feeding for at least 6 months after delivery of a singleton.
Sampling Method: Non-Probability Sample
Enrollment: 394 (Actual)
Dates: Start 2018-06-27 (Actual); Primary Completion 2021-01-14 (Actual); Study Completion 2021-01-14 (Actual)

PRIMARY OUTCOMES:
Proportion of women who are amenorrheic | 6 months postpartum
Proportion of ovulation detected, as measured by serum progesterone levels greater than or equal to 3 ng/mL, in women with a positive urine luteinizing hormone test | 6 months postpartum
Proportion of women who would use the urine luteinizing hormone tests again | 6 months postpartum
  Survey question with responses of yes, no, unsure/maybe

SECONDARY OUTCOMES:
Duration of lactation | within 6 months
Time to resumption of sexual activity | within 6 months
Duration of amenorrhea | within 6 months
Time to initiation of another contraceptive method | within 6 months
Proportion of women who meet criteria for lactational amenorrhea method | at 6 months postpartum
Preliminary estimates of contraceptive efficacy of LAM | within 6 months postpartum
Proportion of women feeding at breast, expressing milk, or both at month 1 postpartum | 1 month postpartum
Proportion of women feeding at breast, expressing milk, or both at month 2 postpartum | 2 months postpartum
Proportion of women feeding at breast, expressing milk, or both at month 3 postpartum | 3 months postpartum
Proportion of women feeding at breast, expressing milk, or both at month 4 postpartum | 4 months postpartum
Proportion of women feeding at breast, expressing milk, or both at month 5 postpartum | 5 months postpartum
Proportion of women feeding at breast, expressing milk, or both at month 6 postpartum | 6 months postpartum
Time to ovulation by method of breastmilk feeding (i.e. primarily breastfeeding or primarily pumping) | within 6 months postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Chen, MD, Principal Investigator — UC Davis
Locations (1):
- University of California, Davis, Sacramento, California, United States